CLINICAL TRIAL: NCT06846944
Title: Mixed-method Research Protocol: Evaluation of a Relaxation Technique for Anxiety Management in Pre-surgical Pediatric Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Gabriella Barresi, Nurse, Meyer Children's Hospital IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LADYBUG
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Surgeries Requiring a Minimum One Day Hospitalization; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ladybug and Sunrise breathing/relaxation technique (Experimental): Ladybug TECHNIQUE is a breathing/relaxation intervention performed in children aged 5 to 10 years and consists of telling the story of a ladybug performing 4 moves and visualizing and performing breathing techniques independently. Afterwards, a drawing is invited.
  SUNRISE TECHNIQUE is a breathing/relaxation intervention performed in children aged 10 to 15 years and consists of having the child imagine a favorite place. Then they are invited to reflect on the experience either verbally or through writing or drawing.
  Interventions: Other: Breathing/relaxation intervention
- Standard of care (No Intervention)

INTERVENTIONS:
Other: Breathing/relaxation intervention — Ladybug TECHNIQUE is a breathing/relaxation intervention performed in children aged 5 to 10 years and consists of telling the story of a ladybug performing 4 moves and visualizing and performing breathing techniques independently. Afterwards, a drawing is invited.
  SUNRISE TECHNIQUE is a breathing/relaxation intervention performed in children aged 10 to 15 years and consists of having the child imagine a favorite place. Then they are invited to reflect on the experience either verbally or through writing or drawing.
  Arms: Ladybug and Sunrise breathing/relaxation technique

SUMMARY:
Children exhibit anxiety before surgery: in particular, the literature reports that younger children have a higher level of preoperative anxiety than older children. Preoperative anxiety has been associated with side effects such as postoperative pain and emergence delirium (ED), which are generally treated with the administration of analgesics but can cause nausea, vomiting, and drowsiness.

In addition to pharmacological strategies, there are behavioral and psychological techniques commonly referred to as nonpharmacological techniques to reduce preoperative anxiety. These are a broad set of strategies and methods, more or less complex, that can be applied to children and adolescents to help them cope with preoperative agitation and for pain control.

Nonpharmacological techniques include distraction techniques that have shown promise in reducing pediatric anxiety and include listening to music , the use of humor, and the use of games . Several researchers have found active distraction to be an effective preoperative anxiolytic in children. Of relevant importance for reducing preoperative anxiety are relaxation techniques as shown in the literature and in particular by a randomized trial that demonstrated the effectiveness of this type of proposed nonpharmacological technique for reducing anxiety and pain in pediatric patients in a preoperative setting.

This study plan to investigate the effectiveness of a breathing/relaxation intervention (Ladybug/Sunshine method) on pediatric patients' anxiety levels before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 years and 15 years;
* Admission for minor surgical conditions of low intensity, such as inguinal hernia, phimosis, sebaceous cysts, vascular malformations, skin lesions, ankyloglossus, afferent to the unified pediatric surgery day-surgery service of AOU Meyer;
* Knowledge of the Italian language and ability to express oneself;

Exclusion Criteria:

* Presence of cognitive impairment reported in history

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage reduction in anxiety score | From recruitment to end of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Meyer Children's Hospital IRCCS, Firenze, Florence, Fi, Italy

IPD SHARING:
Plan to Share IPD: No